CLINICAL TRIAL: NCT00218621
Title: Maternal Buprenorphine Administration and Fetal/Infant Neurobehavior
Brief Title: The Effects of Methadone and Buprenorphine on Fetal Neurobehavior and Infant Neonatal Abstinence Syndrome - 1
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lauren M. Jansson, Associate Professor of Pediatrics Johns Hopkins University School of Medicine, Johns Hopkins University
Other Study IDs: 04032202; R01DA019934 (NIH); NIDA R01DA019934; DPMCDA
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Opiate Dependence; Pregnancy
Keywords: Buprenorphine; Methadone
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Methadone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Buprenorphine / methadone — Parallel study to double blind, double dummy study evaluating safety and efficacy of buprenorphine vs methadone treatment for pregnant opioid dependent women

SUMMARY:
The purpose of this study is to evaluate the effects of drugs used by treatment providers on the fetuses and infants of opiate dependent women. The subjects in this study are women enrolled in a large, multi-site, double blind study that looks at the effects of methadone and buprenorphine treatment during pregnancy. This study will evaluate fetal and maternal biophysiologic data longitudinally during pregnancy to determine how these substances may affect fetal neurobehavior. Additionally, infant neurobehavioral assessments and measurements of infant vagal tone will be collected to see how methadone and buprenorphine differentially affect the neonatal abstinence syndrome, or "withdrawal" in exposed neonates.

DETAILED DESCRIPTION:
Previous research by this group has found that methadone treatment during pregnancy directly impacts fetal neurophysiology independently of maternal physiology. Buprenorphine is a new therapy for opiate dependent individuals, and its use during pregnancy is currently being evaluated. Some research has shown that buprenorphine lessens the neonatal abstinence syndrome when compared to methadone. Thirty methadone and 30 buprenorphine maintained women will be evaluated at 24, 28, 32 and 36 weeks gestation using a state-of-the-art computerized fetal actocardiograph and data analysis program to simultaneously evaluate fetal movement and heart rate and maternal physiologic parameters. Investigators will be blinded to treatment group. Longitudinal neurodevelopment of the fetuses in each group will be explored. The differential effects of methadone and buprenorphine on the neonatal abstinence syndrome will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy opiate dependent women
* currently enrolled in the study "Maternal Opioid Treatment, Human Experimental Research study
* uncomplicated singleton pregnancies

Exclusion Criteria:

* complications of pregnancy, including HIV, diabetes, polyhydramnios, hypertension, preterm labor or placenta previa
* evidence of fetal malformation
* significant maternal health problems, including HIV infection
* significant maternal psychopathology that would preclude informed consent, including schizophrenia
* alcohol dependency per DSM IV criteria

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Opioid dependent pregnant women enrolled in parent study (Maternal Opioid treatment: Human Experimental Research)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Fetal heart rate | up to 300 minutes
Fetal movement | up to 300 minutes

SECONDARY OUTCOMES:
Neonatal abstinence syndrome | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M. Jansson, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Center for Addiction and Pregnancy, Baltimore, Maryland, United States